CLINICAL TRIAL: NCT03101540
Title: Cytokines, PUFA Tissue Concentrations and Treatment Selection in Antenatal MDD
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: William Coryell (Other)
Responsible Party: Sponsor-Investigator, William Coryell, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201102756
Record Dates: First submitted 2017-03-29; First posted 2017-04-05 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder in Pregnancy
Keywords: Major Depressive Disorder,; omega-3 polyunsaturated fatty acid; PUFA; Pregnancy; eicosapentaenoic acid (EPA) supplementation; cytokine; docosahexaenoic acid (DHA)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Eicosapentaenoic Acid; Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: A single group model was used: pregnant women.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supplementation (Experimental): Subjects received Omega-3 PUFA supplementation
  Interventions: Drug: Omega-3 PUFA supplementation

INTERVENTIONS:
Drug: Omega-3 PUFA supplementation — Subjects received 2.2g of eicosapentaenoic acid (EPA) and 1.2g of docosahexaenoic acid (DHA) daily for the duration of the study.
  Other Names: eicosapentaenoic acid (EPA); docosahexaenoic acid (DHA)

SUMMARY:
For a number of reasons women with major depressive disorder often discontinue conventional antidepressants when they become pregnant and prefer not to take them when depressive illness develops in the course of pregnancy. There is now considerable evidence that the administration of the omega-3 polyunsaturated fatty acid, eicosapentaenoic acid (EPA), as monotherapy has antidepressant effects. If it could be clearly established as effective such an approach would offer a valuable alternative for woman who are at risk for, or who develop, depressive disorder during pregnancy. Strongly positive placebo-controlled trials of EPA supplementation, though, co-exist with entirely negative ones. No clear reasons for these discrepancies have emerged but one possibility is that the samples studied have differed in the proportion of individuals likely to benefit from EPA supplementation. As there has been no effort to identify such individuals we propose to explore two groups of measures, both relevant to EPA's likely mechanisms of action, as potential tools for identifying individuals likely to benefit this treatment. Hypothesis: Among women who experience major depressive episodes during their first two trimesters of pregnancy, baseline measures of cytokine activity and erythrocyte PUFA concentrations will be associated, in an additive or interactive fashion, with subsequent improvement in depressive symptoms among women taking omega-3 PUFA supplementation.

DETAILED DESCRIPTION:
This is a project to determine whether certain measures of nutritional status and immune functioning can be useful in the identification of women who would most benefit from omega-3 supplements as treatment for depression during pregnancy.

Pregnancy does not reduce the risk of recurrence among women who have previously experienced depressive illness and the advent of new episodes during pregnancy raises particular problems. Concerns over the possible teratogenicity of medications in general leave many women reluctant to continue preexisting antidepressant prophylaxis or to accept new trials of conventional antidepressant treatment and there is accumulating evidence that the SSRIs have short-term adverse effects on the newborn. The antidepressant effects of omega-3 polyunsaturated fatty acid (PUFA) supplementation may offer a particularly appropriate alternative to conventional therapy for depressive episodes that occur during pregnancy. The nutritional needs of the fetus increase the likelihood of omega-3 PUFA deficits in the mother but access to adequate omega-3 PUFAs but fish intake is limited due to concerns over mercury levels. Antidepressant trials of omega-3 supplementation that have described significant benefits over placebo include one that targeted pregnant women and yielded a large effect size. Other trials, however, have failed to show clear antidepressant effects and meta-analyses have yielded no explanations for these inconsistencies. A clear possibility is that the studies with positive results involved subjects who more likely to benefit from omega-3 supplementation but the characteristics of such individuals are entirely unknown. Numerous case-control studies have associated depressive illness with lower tissue concentration of omega-3 PUFAs and with higher ratios of omega-6 to omega-3. Such measures may well identify individuals likely show antidepressant effects from supplementation. The likelihood that omega-3 PUFAs exert antidepressant effects via modulation of the inflammatory cascade, and the extensive evidence that high levels of cytokines characterize individuals with depressive disorders, indicate that these measures too may help to select those most likely to benefit from treatment with omega-3 PUFAs. A group of 60 women who begin pregnancy in depressive episodes or who develop episodes in their first two trimesters but who choose not to take conventional antidepressant therapy would be used to test PUFA tissue concentration and inflammatory measures as predictors of response to omega-3 supplementation monotherapy. Aim #1: To determine, among women with first- or second-trimester major depressive episodes, relationships between subsequent response to omega-3 PUFA supplementation and baseline measures of PUFA erythrocyte concentrations and cytokine activity.

Hypothesis #1: Among women who experience major depressive episodes during their first two trimesters of pregnancy, baseline measures of cytokine activity and erythrocyte PUFA concentrations will be associated, in an additive or interactive fashion, with subsequent improvement in depressive symptoms among women taking omega-3 PUFA supplementation. Aim #1 will test whether measures of PUFA tissue concentrations and cytokine activity have potential value in treatment selection for women who experience depressive disorder during pregnancy. The strength with which measures correlate with symptom outcome will be used to select those for use in a definitive placebo-controlled trial that will target a sample enriched for those likely to respond to EPA supplementation.The measures that emerge most strongly as risk factors for new episodes would then be used to select subjects for participation in a placebo-controlled trial of EPA supplementation as prophylaxis against depressive disorder recurrence. The results would be integrated into the design of both acute treatment and prophylaxis trials.

ELIGIBILITY:
Inclusion Criteria:

1. women with uncomplicated pregnancies and within 24 weeks of their last menstrual period
2. describe symptoms over the previous two weeks sufficient to meet DSM IV criteria for MDD as determined by the SCID
3. have a 21-item HAM-D of 16 or more

Exclusion Criteria:

1. antidepressant use in preceding month
2. use in previous 2 wks of non-steroidal anti-inflammatory drugs (NSAIDS), antibiotics or glucocorticoids
3. use in previous 2 wks of psychotropic medications other than hypnotics or benzodiazepines in diazepam dose-equivalents greater than 2mg/day for insomnia
4. a previous diagnosis of an autoimmune disease, of hyperlipidemia, or of schizophrenia or schizoaffective disorder
5. evidence of substance dependence in previous 6 months
6. preoccupation with, or plans for, suicide
7. a history of hypersensitivity to fish or fish oil supplements
8. current use of anticoagulants
9. any current medical condition associated with clinically significant decreases in coagulability, i.e. systemic lupus erythematosis, VonWillebrend's disease
10. the initiation of regularly scheduled course of psychotherapy within the previous 2 months
11. current use of category D or category X medications

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study is focused on pregnant women.
Enrollment: 27 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HAM-D) | Subjects were administered the HAM-D at Day 1 and every month thereafter until week 38 of their pregnancies. At 2 months postpartum it was again administered by phone.
  The HAM-D is a multiple item semi-structured clinician administered questionnaire used to assess the range, type and severity of depressive symptoms observed in patients with MDD. The HAM-D24 consists of 24 symptoms, each of which is rated from 0 to 2 or 0 to 4, where 0 is none/absent. The HAMD-24 total score is calculated as the sum of the 24 individual symptom scores; the total score can range from 0 to 76. Higher HAMD-24 scores indicate more severe depression.
Montgomery-Asberg Depression Scale (MADRS) | Subjects were administered the MADRS on Day 1 and every month thereafter until week 38 of their pregnancies. At 2 months postpartum e ach subject was again administered the MADRS by phone.
  The MADRS is a clinician administered semi-structured scaled designed to detect changes in depressive symptoms. The scale contains 10 items and ratings are graded from 0 to 6 , with 0 representing an absence of a symptom and 6 corresponding to the most severe degree of MDD symptomology.
Edinburgh Postnatal Depression Scale (EPDS) | Subjects were asked to complete the EPDS on Day 1 and every month thereafter until week 38 of their pregnancies and then again 2 months postpartum by phone.
  The EPDS is a self-administered depression screen for postpartum women. The EPDS consists of 10 questions. Responses are scored 0,, 1, 2, or 3 according to increased severity of the symptom. Items marked with an * are reversed scored. A total score of 13 or more suggests follow-up intervention is warranted.
Beck Depression Scale (BDI) | Subjects were asked to complete the BDI on Day 1 and every month thereafter through week 38 of their pregnancies and then again 2 months postpartum by phone.
  The BDI is a self-administered questionnaire developed to detect, assess, and monitor changes in depressive symptoms. It is composed of 21 items, each with 4 possible responses scored from 0 to 3 with 3 indicating a higher level of severity. For people who have been clinically diagnosed, scores from 0 to 9 represent minimal depressive symptoms, scores of 10 to 16 indicate mild depression, scores of 17 to 29 indicate moderate depression, and scores of 30 to 63 indicate severe depression.

IPD SHARING:
Plan to Share IPD: No
The Investigator will not be sharing IPD

REFERENCES:
- [Background] Hibbeln JR. Seafood consumption, the DHA content of mothers' milk and prevalence rates of postpartum depression: a cross-national, ecological analysis. J Affect Disord. 2002 May;69(1-3):15-29. doi: 10.1016/s0165-0327(01)00374-3. PMID 12103448
- [Background] De Vriese SR, Christophe AB, Maes M. Lowered serum n-3 polyunsaturated fatty acid (PUFA) levels predict the occurrence of postpartum depression: further evidence that lowered n-PUFAs are related to major depression. Life Sci. 2003 Nov 7;73(25):3181-7. doi: 10.1016/j.lfs.2003.02.001. PMID 14561523
- [Background] Peet M, Murphy B, Shay J, Horrobin D. Depletion of omega-3 fatty acid levels in red blood cell membranes of depressive patients. Biol Psychiatry. 1998 Mar 1;43(5):315-9. doi: 10.1016/s0006-3223(97)00206-0. PMID 9513745
- [Background] Rees AM, Austin MP, Owen C, Parker G. Omega-3 deficiency associated with perinatal depression: case control study. Psychiatry Res. 2009 Apr 30;166(2-3):254-9. doi: 10.1016/j.psychres.2007.12.011. Epub 2009 Mar 5. PMID 19268372